CLINICAL TRIAL: NCT06471621
Title: PrEcision Medicine in the Management of Cardiovascular Surgery Associated AKI - PEAK: a Prospective Observational Cohort Study
Brief Title: Precision Medicine in Cardiovascular Surgery Associated Acute Kidney Injury
Acronym: PEAK
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: CSL Behring (Industry)
Responsible Party: Sponsor
Other Study IDs: DLF-Nr: 5658; BASEC-Nr: 2023-02024 (Other: swissethics)
Record Dates: First submitted 2024-04-24; First posted 2024-06-24 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Acute Kidney Injury; Surgery-Complications; Frailty
Keywords: Kidney; Renal; Cardiac; Thoracic; Abdominal; Valvular replacement; CABG; Aneurysm; cardiopulmonary bypass; Ischemia
MeSH Terms: conditions — Acute Kidney Injury; Frailty; Aneurysm; Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, Plasma, Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this prospective observational study is to define a risk profile for cardiovascular surgery associated acute kidney injury (AKI), using clinical patient characteristics, operation parameters as well as blood and urine laboratory values.

The main question it aims to answer is:

• Does a combination of the factors mentioned above better predict patient outcome than classical factors used to date in clinical practice?

Participants of this study are adults aged 18 and above who are scheduled for elective heart or main artery surgery, and who have given written informed consent.

DETAILED DESCRIPTION:
The difficulty of precisely predicting AKI following major surgery is a clinical challenge and unmet need as treatment should be introduced within 24-48 hours. In addition there is no available treatment to date apart from supportive therapy such as renal replacement therapy.

Therefore, early identification of patient-specific biomarkers and other clinical predictors could help to better understand the association with AKI and other patient outcomes. In addition to the "classical" risk factors (age, diabetes, pre-existing CKD), frailty might represent another important variable, as shown in previous observational studies. Importantly frailty is not unique to age, although it occurs in approximately 25% of those over 65 and affects more than half of the population aged 85 and older, as it has been shown to be highly prevalent in hospitalized patients and/or patients with CKD. Furthermore, in preclinical studies the serum protein Fetuin-A was identified as potential biomarker for vascular surgery associated AKI.

PEAK is a single center, prospective observational study involving several clinics at the University Hospital Bern. Besides from demographic data and perioperative parameters, blood and urine are collected with high granularity during and immediately after surgery (15min after the first cut, start and end of cardiopulmonary bypass (CBP) or aortic clamping (X-clamp), 4 hours after surgery) and at day 1, 2, 3, and 7 (or discharge) post-surgery. In addition renal function will be assessed at day 90. Furthermore, study participants will answer the Edmonton frailty questionnaire at baseline and at day 90.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective cardiovascular surgery, such as valvular replacement surgery, with or without combined coronary artery bypass graft (CABG), or thoracic or abdominal aortic surgery.
* Written informed consent obtained prior to surgery.

Exclusion Criteria:

* Patients with a kidney transplant or on renal replacement therapy
* Severe liver failure, defined by the presence of encephalopathy, Factor V < 50% and INR >1.5 on preoperative blood sample (within 4 weeks).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective cardiovascular surgery at the University Hospital Bern (Inselspital), Switzerland
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-06-16 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of serum Fetuin-A values | Baseline to day 90
  Measurement of serum Fetuin-A at baseline and at the various sampling time-points mentioned above.

SECONDARY OUTCOMES:
BMI | Baseline and day 90
  Body mass index of participants in (kg/m2), integer: min 15 (extreme underweight), max 45 (extreme overweight)
eGFR | Baseline and day 90
  estimated glomerular filtration rate in (ml/min)
Proteinuria | Baseline and day 90
  Albumin in urine normalized to creatinine in categorized into 3 groups:
  1. <30 mg/d
  2. 30-300 mg/d
  3. >300 mg/d
ASA score | Baseline
  American Society of Anesthesiology classification of physical status (1-6)
  1. - Normal health
  2. - Mild systemic disease
  3. - Severe systemic disease
  4. - Severe systemic disease that is constant threat to life
  5. - Moribund, not expected to survive 24h with or without operation
  6. - Declared brain-dead
Euroscore II | Baseline
  Euroscore II, predicted mortality in (%)
STS score (only for cardiac surgery) | Baseline
  Society of Thoracic Surgeons Score in (%), higher values predict higher risk
Duration of ECC (only for cardiac surgery) | Peri-operative
  Time on extracorporeal circuit in (min)
Duration of X-clamp (only for aortic surgery) | Peri-operative
  Time of X-clamping in (min)
Lowest body temperature | Peri-operative
  Lowest body temperature recorded during surgery in (°C)
SAPS II score | After Operation to day 7
  Simplified Acute Physiology Score (SAPS) II°C), in-hospital mortality at ICU admission, integer min 1, max 200, higher values predict higher mortality
Urine output | After Operation to day 7
  Daily urine volume in (ml)
Assessment of AKI incidence and severity at day 7 in association with change in serum Fetuin-A levels over time | Baseline to day 7
  AKI will be assessed as a binary outcome (presence/absence)
  Biomarkers for AKI severity include levels of direct Fetuin-A targets, kidney function parameters, predictors of AKI or CKD (NGAL, suPAR, Nephrocheck®, or YKL-40), hemolysis (hemoglobin, transferrin), inflammatory mediators (cytokines, chemokines or growth factors), and exploratory assessments (proteomics, metabolomics).
Assessment of AKI to CKD progression at day 90 in association with change in serum Fetuin-A levels over time | Baseline to day 90
  CKD will be evaluated as a binary outcome (presence/absence) based on renal functional parameters.
Assessment of the patient-reported outcome measure (PROM) frailty in association with progression to CKD and worse clinical outcome | Baseline and day 90
  Frailty in terms of patient-related outcome will be reported as a paired difference of mean frailty score (Edmonton Frail Scale) between baseline and 90-days visit. The scale ranges from 0 (not frail) to 17 (severe frailty).
Grip strength | Baseline and day 90
  Grip strength of dominant hand in kg

CONTACTS AND LOCATIONS:
Overall Officials: Uyen Huynh-Do, Prof. MD, Principal Investigator — University Hospital Bern (Inselspital)
Locations (1):
- University Hospital Bern (Inselspital), Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hammer N, Rudloff S, Waskowski J, Pfortmuller C, Pingpoh C, Chaikhouni B, Herzig S, Rheinberger M, Pedersen E, Luder G, Kotelis D, Siepe M, Erdoes G, Schefold J, Huynh-Do U. Protocol of the exploratory prospective observational PEAK study: PrEcision medicine in the management of cardiovascular surgery associated Acute Kidney Injury (AKI). BMJ Open. 2025 Jul 30;15(7):e095817. doi: 10.1136/bmjopen-2024-095817. PMID 40744512